CLINICAL TRIAL: NCT03405259
Title: A Pilot Clinical Study to Compare Professional Treatments for Dentinal Hypersensitivity
Brief Title: A Clinical Study to Compare Professional Treatments for Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013077
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Dentinal Hypersensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Super Seal® Desensitizer (Experimental): Professionally Applied
  Interventions: Device: Super Seal® Desensitizer
- Acclean® Fluoride Varnish (Sham Comparator): Professionally Applied
  Interventions: Device: Acclean® Fluoride Varnish

INTERVENTIONS:
Device: Super Seal® Desensitizer — Single dose professional application.
  Arms: Super Seal® Desensitizer
Device: Acclean® Fluoride Varnish — Single dose professional application.
  Arms: Acclean® Fluoride Varnish

SUMMARY:
The objective of this study is to compare professional treatments for dentinal hypersensitivity immediately following a single, professionally-applied treatment and again approximately 2 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* be in good general health as determined by the Investigator/designee; and
* have at least one tooth with a VAS score of greater than or equal to 30 in response to the air challenge.

Exclusion Criteria:

* allergy to rosin or to pine nuts;
* self-reported pregnancy or nursing;
* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* active treatment for periodontitis;
* fixed facial orthodontic appliances;
* any diseases or conditions that might interfere with the safe completion of the study; or
* an inability to undergo any study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2013-09-13 (Actual); Study Completion 2013-09-13 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Super Seal® Desensitizer | Acclean® Fluoride Varnish
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Super Seal® Desensitizer | Acclean® Fluoride Varnish | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.84) | 48.1 (19.71) | 46.4 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Oriental | 1 | 1 | 2
  Black | 0 | 1 | 1
  Caucasian | 8 | 9 | 17
  Hispanic | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A negative change from Baseline score represents a decrease in sensitivity from baseline.The mean change from Baseline was calculated for this measure.
Time Frame: Within 5 minutes after treatment was applied
Population: Twenty-two (22) subjects received study product and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Super Seal® Desensitizer | Acclean® Fluoride Varnish
Number analyzed (Participants) | 11 | 11
Units on a scale | -0.55 (0.69) | -0.95 (0.93)

2. Primary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced. A negative change from Baseline score represents a decrease in sensitivity from baseline.
Time Frame: Within 5 minutes after treatment was applied
Population: Twenty-two (22) subjects received product and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Super Seal® Desensitizer | Acclean® Fluoride Varnish
Number analyzed (Participants) | 11 | 11
Units on a scale | -17.60 (21.32) | -19.55 (25.15)

ADVERSE EVENTS:
Arm/Group | Super Seal® Desensitizer | Acclean® Fluoride Varnish
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other